CLINICAL TRIAL: NCT01047306
Title: A Longitudinal, Prospective, Natural History Study of Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Brief Title: A Study of Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-SAN-053
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Sanfilippo Syndrome Type A
MeSH Terms: conditions — Mucopolysaccharidosis III | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF, urine and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment: This is a longitudinal, prospective, observational, natural history study of patients with MPS IIIA to identify potential surrogate endpoints for future ERT trials via standardized clinical, biochemical, neurocognitive, developmental, behavioral and imaging measures.
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — Physical, developmental, neurological, behavioral, and neurocognitive assessments

SUMMARY:
The purpose is to evaluate the course of disease progression in MPS IIIA patients who are untreated to identify potential surrogate endpoints that may be utilized in future ERT trials of MPS IIIA via defined assessments including standardized clinical, biochemical, neurocognitive, behavioral, developmental, and imaging measures.

ELIGIBILITY:
Inclusion Criteria:

1a. Documented deficiency in HNS enzyme activity of less than or equal to 10% of the lower limit of the normal range as measured in fibroblasts or leukocytes (based on normal range for diagnosis of MPS IIIA by a laboratory that is acceptable to Shire HGT).

AND

1b. Normal enzyme activity level of at least one other sulfatase (to rule out multiple sulfatase deficiency) as measured in fibroblasts or leukocytes (based on normal range by a laboratory that is acceptable to Shire HGT).

2.Patient is greater than or equal to 1 year of age and developmental age greater than or equal to 1 year.

3. Patient is medically stable to accommodate the protocol requirements, including travel and assessments, without placing an undue burden on the patient/patient's family.

4. Voluntarily signed an IRB/IEC-approved informed consent (assent if applicable) form. The patient's, patient's parents or legally authorized representative(s) consent and patient's assent as appropriate, must be obtained.

Exclusion Criteria:

1. Patient has significant non-MPS IIIA-related CNS impairment or behavioral disturbances, which would confound the scientific integrity or interpretation of study assessments, as determined by the investigator.
2. Patients who, for MPS IIIA behavioral-related reasons,in the opinion of the investigator, would preclude performance of study neurocognitive and developmental testing procedures.
3. Patients who are pregnant, breast feeding, or female patients of childbearing potential, who will not or cannot comply with the use of an acceptable method of birth control such as condoms, barrier method, oral contraception, etc.
4. Patient is blind and/or deaf.
5. Patient has any known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptably high risk for anesthesia due to airway compromise or other conditions.
6. Patient or patient family history of neuroleptic malignant syndrome, malignant hyperthermia, or other anesthesia-related concerns.
7. The Investigator may choose to exclude patients who have had complications resulting from prior lumbar punctures.
8. Patient history of poorly controlled seizure disorder.
9. Patient history of an intracranial pressure (ICP) or opening CSF pressure upon lumbar puncture that exceeds 30 cm water that has not been definitively treated.
10. Patient is currently receiving psychotropic or other medications which in the investigator's opinion, would be likely to substantially confound test results.
11. Patient cannot sustain absence from aspirin, non-steroidals, or medications that affect blood clotting within 1 week prior to a relevant study related procedure (eg, lumbar puncture if applicable), or has ingested such medications within 1 week before any procedures in which any change in clotting activity would be deleterious.
12. Patient has received treatment with any investigational drug or device intended as a treatment for MPS IIIA within the 30 days prior to, or during the study, or is currently enrolled in another study that involves an investigational drug or device (enrollment through Safety follow-up contact).
13. Patient has received a hematopoietic stem cell or bone marrow transplant.
14. Patient's assent is unattainable, or the patient's parent(s), or patient's legally authorized representative(s) is/are unable to understand the nature, scope, and possible consequences of the study, or do/does not agree to comply with the protocol defined schedule of assessments.
15. The patient has any item (braces, tattoos, etc.) which would exclude the patient from being able to undergo MRI according to local Institutional Policy, or the patient has any other situation that would exclude the patient from undergoing any other procedure required in this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Initial patient eligibility is based on patient age and on a confirmed diagnosis of MPS IIIA by biochemical enzyme assay.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-02-15 (Actual); Primary Completion 2013-07-10 (Actual); Study Completion 2013-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cingi EC, Beebe DS, Whitley CB, Belani KG. Anesthetic care and perioperative complications in children with Sanfilipo Syndrome Type A. Paediatr Anaesth. 2016 May;26(5):531-8. doi: 10.1111/pan.12876. Epub 2016 Mar 9. PMID 26956723
- [Derived] Shapiro EG, Nestrasil I, Delaney KA, Rudser K, Kovac V, Nair N, Richard CW 3rd, Haslett P, Whitley CB. A Prospective Natural History Study of Mucopolysaccharidosis Type IIIA. J Pediatr. 2016 Mar;170:278-87.e1-4. doi: 10.1016/j.jpeds.2015.11.079. Epub 2016 Jan 16. PMID 26787381
- [Derived] Shapiro EG, Nestrasil I, Ahmed A, Wey A, Rudser KR, Delaney KA, Rumsey RK, Haslett PA, Whitley CB, Potegal M. Quantifying behaviors of children with Sanfilippo syndrome: the Sanfilippo Behavior Rating Scale. Mol Genet Metab. 2015 Apr;114(4):594-8. doi: 10.1016/j.ymgme.2015.02.008. Epub 2015 Mar 5. PMID 25770355
- [Derived] Rumsey RK, Rudser K, Delaney K, Potegal M, Whitley CB, Shapiro E. Acquired autistic behaviors in children with mucopolysaccharidosis type IIIA. J Pediatr. 2014 May;164(5):1147-1151.e1. doi: 10.1016/j.jpeds.2014.01.007. Epub 2014 Feb 25. PMID 24582005

RESULTS

PARTICIPANT FLOW:
Groups:
- Children < 6 Years Old: Children ≥1 to < 6 years of age with Sanfilippo Syndrome Type A (mucopolysaccharidosis type IIIA; MPS IIIA) who were untreated with any investigational products (drugs and/or devices).
- Children ≥ 6 Years Old: Children ≥ 6 years of age with Sanfilippo Syndrome Type A (mucopolysaccharidosis type IIIA; MPS IIIA) who were untreated with any investigational products (drugs and/or devices).
Period: Overall Study
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Started | 19 | 6
Discontinued From the Study | 3 | 0
Completed | 16 | 6
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: A maximum of 25 patients with MPS IIIA will be enrolled in the study to provide at least 12 patients who complete the study. This number was not based on any statistical consideration, but is expected to be adequate to describe the natural progression of Sanfilippo A syndrome.
Groups:
- Children < 6 Years Old: Children ≥1 to < 6 years of age with MPS IIIA who were untreated with any investigational products (drugs and/or devices).
- Children ≥ 6 Years Old: Children ≥ 6 years of age with MPS IIIA who were untreated with any investigational products (drugs and/or devices).
- Total: Total of all reporting groups
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old | Total
Number analyzed (Participants) | 19 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.29 (1.996) | 12.44 (4.500) | 6.24 (4.452)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 13 | 3 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bayley Scales of Infant Development-III/Kaufman Assessment Battery for Children-II (BSID-III/KABC-II) Age-Equivalent Scores
Description: Children 1 year-42 months were assessed by the BSID-III; those >42 months and with a developmental age of >42 months by the Vineland Adaptive Behavior Scales-II (VABS-II) were evaluated with the KABC-II. For children >42 months, but <42 months in developmental age, and those unable to complete at least 3 cognitive KABC-II subtests, the BSID-III was used. The BSID-III is a series of measurements to assess the motor, language, and cognitive development of infants and toddlers and consists of a series of developmental play tasks. The KABC-II is an individually administered measure of processing/reasoning abilities. Raw scores were converted to age- equivalent scores to measure ability, skill, and knowledge, expressed as the age at which most individuals reach the same level (age norm; range: 0, unbound ). A positive value indicates improvement. The BSID-III and KABC-II age- equivalent scores were based on the cognitive domain and average non-verbal age-equivalent score, respectively.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: All analyses were based on the Main Analysis Population, which included all enrolled patients. Data were not available for all patients at all time points.
Measure: Mean (Standard Deviation); unit: months
Groups:
- Children < 6 Years: Children ≥1 to < 6 years of age with MPS IIIA who were untreated with any investigational products (drugs and/or devices).
- Children ≥ 6 Years: Children ≥ 6 years of age with MPS IIIA who were untreated with any investigational products (drugs and/or devices).
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
months
  6 months, n=18,6 | 0.17 (2.093) | 1.19 (3.289)
  12 months, n=18,6 | -1.72 (4.625) | 1.39 (4.029)
  End of Study, n=15,5 | -1.80 (7.143) | 2.95 (4.652)

2. Primary Outcome: Change From Baseline in BSID-III/KABC-II Developmental Quotient (DQ) Scores
Description: The determination of whether a patient received BSID-III was based on an algorithm that includes the patient's calendar age and VABS-II age -equivalent score (See Outcome 1). The BSID-III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. The KABC-II is an individually administered measure of processing and reasoning abilities. The DQ is a means to express a neurodevelopmental/cognitive delay. The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range: 0, 100). The BSID-III DQ score is based on the cognitive domain. The DQ score for KABC-II is calculated from the average non-verbal age-equivalent score. A positive value indicates improvement in health and cognition.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of chronological age
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
percentage of chronological age
  6 months, n=18,6 | -7.42 (6.153) | -0.03 (1.960)
  12 months, n=18,6 | -15.69 (9.258) | -1.66 (2.977)
  End of Study, n=15,5 | -26.09 (14.788) | -2.94 (2.588)

3. Primary Outcome: Change From Baseline in Vineland Adaptive Behavior Scales-II (VABS-II) Age-equivalent Scores
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. It is an instrument that supports the diagnosis of intellectual and developmental disabilities in patients from birth to 90 years. This test measures the following 5 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). The mean age-equivalent score is obtained by averaging out the age-equivalent scores for the all the sub-domains except for Gross and Fine motor skills (range: 0, unbound). A positive value indicates improvement in health and cognition
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
months
  6 months, n=17,6 | -0.92 (3.966) | -1.11 (5.661)
  12 months, n=18,6 | -0.90 (8.170) | -2.63 (4.847)
  End of Study, n=16,6 | -2.29 (8.321) | -7.80 (15.834)

4. Primary Outcome: Change From Baseline in VABS-II Overall DQ Scores
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. It is an instrument that supports the diagnosis of intellectual and developmental disabilities in patients from birth to 90 years. This test measures the following 5 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). The DQ is a means to express a neurodevelopmental/cognitive delay. The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range, 0, 100). The overall DQ score is calculated from the mean age-equivalent score obtained by averaging out the age-equivalent scores for the all the sub-domains except for Gross and Fine motor skills. A positive value indicates improvement in health and cognition.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of chronological age
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
percentage of chronological age
  6 months, n=17,6 | -9.33 (8.632) | -2.78 (5.971)
  12 months, n=18,6 | -12.88 (15.131) | -5.12 (7.683)
  End of Study, n=16,6 | -23.81 (14.655) | -9.70 (11.299)

5. Other Pre Specified Outcome: Change From Baseline in Urine Glycosaminoglycan (GAG) Levels
Description: Urine GAG was measured by a dye binding assay. A negative value indicates that GAG levels decreased.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg GAG/mmol creatinine
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
mg GAG/mmol creatinine
  6 months, n=18,6 | 0.26 (19.379) | -10.23 (32.983)
  12 months, n=18,6 | -0.39 (19.429) | -7.95 (31.516)
  End of Study, n=15,5 | -0.33 (22.706) | -6.34 (28.810)

6. Secondary Outcome: Change From Baseline Values in Gray Matter Volume Assessed by Brain Magnetic Resonance Imaging (MRI)
Description: Total brain cortical gray matter volume was determined by analysis of brain MRI. The analysis was performed using "Freesurfer" software, which provides completely automated parcellation of the brain cortex and subcortical structures. In some cases, manual adjustments were necessary in cases of intensity normalization failure, resulting in erroneous white matter segmentation. A negative value indicates that gray matter volume decreased.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
milliliters
  6 months, n=17,6 | -15.98 (21.860) | 1.16 (14.790)
  12 months, n=16,6 | -41.40 (36.319) | -11.68 (13.126)
  End of Study, n=9,5 | -80.29 (45.867) | -22.41 (18.134)

7. Secondary Outcome: Change From Baseline in The Total Disability Score (TDS) of The Four Point Scoring System (FPSS)
Description: The FPSS is an MPS III-specific disability assessment that evaluates motor function, expressive language, and cognitive function on a 0- to 3- point scale and can be used for individuals of all ages. A score of 3 points is assigned for normal function, 2 points for beginning of regression, 1 point for severe level of regression, and 0 points for lost skills. The total disability score (TDS) is the average of the motor function, speech, and cognitive function scores (range: 0, 3). The scoring is based on the parent's response to a detailed questionnaire that covers several aspects of the disease. A positive value indicates improvement in function.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
units on a scale
  6 months, n=18,6 | -0.18 (0.411) | 0.10 (0.245)
  12 months, n=18,6 | -0.31 (0.512) | 0.10 (0.245)
  End of Study, n=15,5 | -0.43 (0.448) | 0.18 (0.164)

8. Secondary Outcome: Percent of Participants With an Abnormal Overall Test Result of Auditory Brainstem Response (ABR) at Baseline
Description: Hearing loss in subjects with MPS IIIA was characterized by assessing the ABR. The ABR is a voltage response evoked by acoustic stimuli as sound is processed along the auditory pathway. It consists of electrical signals resulting from the sum of sound-evoked activity along the auditory nerve and brainstem nuclei. The ABR analysis determines the sound intensity at which a neural response first appears (hearing threshold). Other parameters of interest include amplitude (the number of neurons firing), latency (the speed of transmission), interpeak latency (the time between peaks), and interaural latency (the difference in wave V latency between ears). The interpeak latency I-V interval (or central transmission time) is considered the most reliable index of brainstem function. Auditory brainstem response assessments were conducted under anesthesia. An abnormal value was greater than 21 decibels hearing level (dBHL).
Time Frame: Baseline
Population: All analyses were based on the Main Analysis Population, which included all enrolled patients. Data were not available for all patients.
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=11,5 | 57.9 | 50.0
  Left ear, n=11,5 | 57.9 | 66.7

9. Secondary Outcome: Percent of Participants With an Abnormal Overall Test Result of Auditory Brainstem Response (ABR) at 6 Months
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=18,6 | 94.7 | 66.7
  Left ear, n=18,6 | 94.7 | 66.7

10. Secondary Outcome: Percent of Participants With an Abnormal Overall Test Result of Auditory Brainstem Response (ABR) at 12 Months
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=17,6 | 89.5 | 66.7
  Left ear, n=17,6 | 89.5 | 83.3

11. Secondary Outcome: Percent of Participants With an Abnormal Overall Test Result of Auditory Brainstem Response (ABR) at End of Study
Description: as for outcome 8
Time Frame: End of Study (12 months assessment or early termination)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=15,5 | 73.7 | 66.7
  Left ear, n=15,5 | 78.9 | 66.7

12. Secondary Outcome: Percent of Participants With Sensorineural Hearing Loss at Baseline, as Assessed by the Auditory Brainstem Response (ABR)
Description: Sensorineural hearing loss occurs from damage to the inner ear, the brain, or the nerve that runs from the ear to the brain (auditory nerve). Hearing loss in subjects with MPS IIIA was characterized by assessing the ABR. The ABR is a voltage response evoked by acoustic stimuli as sound is processed along the auditory pathway. It consists of electrical signals resulting from the sum of sound-evoked activity along the auditory nerve and brainstem nuclei. The ABR analysis determines the sound intensity at which a neural response first appears (hearing threshold). Other parameters of interest include amplitude (the number of neurons firing), latency (the speed of transmission), interpeak latency (the time between peaks), and interaural latency (the difference in wave V latency between ears). The interpeak latency I-V interval (or central transmission time) is considered the most reliable index of brainstem function. Auditory brainstem response assessments were conducted under anesthesia.
Time Frame: Baseline
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=9,3 | 21.1 | 16.7
  Left ear, n=9,4 | 21.1 | 16.7

13. Secondary Outcome: Percent of Participants With Sensorineural Hearing Loss at 6 Months, as Assessed by the Auditory Brainstem Response (ABR)
Description: as for outcome 12
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=18,4 | 63.2 | 50.0
  Left ear, n=18,4 | 57.9 | 50.0

14. Secondary Outcome: Percent of Participants With Sensorineural Hearing Loss at 12 Months, as Assessed by the Auditory Brainstem Response (ABR)
Description: as for outcome 12
Time Frame: 12 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=17,4 | 84.2 | 50.0
  Left ear, n=17,5 | 89.5 | 50.0

15. Secondary Outcome: Percent of Participants With Sensorineural Hearing Loss at End of Study, as Assessed by the Auditory Brainstem Response (ABR)
Description: as for outcome 12
Time Frame: End of Study (12 months assessment or early termination)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=14,4 | 68.4 | 66.7
  Left ear, n=15,4 | 78.9 | 66.7

16. Secondary Outcome: Percent of Participants With Conductive Hearing Loss at Baseline, as Assessed by the Auditory Brainstem Response (ABR)
Description: Conductive hearing loss occurs when there is a problem conducting sound waves along the route through the outer ear, tympanic membrane, or middle ear. Hearing loss in subjects with MPS IIIA was characterized by assessing the ABR. The ABR is a voltage response evoked by acoustic stimuli as sound is processed along the auditory pathway. It consists of electrical signals resulting from the sum of sound-evoked activity along the auditory nerve and brainstem nuclei. The ABR analysis determines the sound intensity at which a neural response first appears (hearing threshold). Other parameters of interest include amplitude (number of neurons firing), latency (speed of transmission), interpeak latency (time between peaks), and interaural latency (difference in wave V latency between ears). The interpeak latency I-V interval (or central transmission time) is considered the most reliable index of brainstem function. Auditory brainstem response assessments were conducted under anesthesia.
Time Frame: Baseline
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=9,3 | 10.5 | 0.0
  Left ear, n=9,4 | 10.5 | 16.7

17. Secondary Outcome: Percent of Participants With Conductive Hearing Loss at 6 Months, as Assessed by the Auditory Brainstem Response (ABR)
Description: as for outcome 16
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=18,4 | 5.3 | 0.0
  Left ear, n=18,4 | 5.3 | 0.0

18. Secondary Outcome: Percent of Participants With Conductive Hearing Loss at 12 Months, as Assessed by the Auditory Brainstem Response (ABR)
Description: as for outcome 16
Time Frame: 12 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=17,4 | 0.0 | 0.0
  Left ear, n=17,5 | 0.0 | 16.7

19. Secondary Outcome: Percent of Participants With Conductive Hearing Loss at End of Study, as Assessed by the Auditory Brainstem Response (ABR)
Description: as for outcome 16
Time Frame: End of Study (12 months assessment or early termination)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Right ear, n=14,4 | 0.0 | 0.0
  Left ear, n=15,4 | 0.0 | 0.0

20. Secondary Outcome: Number of Participants With Mild, Moderate, or Severe Hearing Loss at Baseline, as Assessed by The Auditory Brain Response (ABR)
Description: Hearing loss in subjects with MPS IIIA was characterized by assessing the ABR. The ABR is a voltage response evoked by acoustic stimuli as sound is processed along the auditory pathway. It consists of electrical signals resulting from the sum of sound-evoked activity along the auditory nerve and brainstem nuclei. The ABR analysis determines the sound intensity at which a neural response first appears (hearing threshold). Other parameters of interest include amplitude (the number of neurons firing), latency (the speed of transmission), interpeak latency (the time between peaks), and interaural latency (the difference in wave V latency between ears). The interpeak latency I-V interval (or central transmission time) is considered the most reliable index of brainstem function. Auditory brainstem response assessments were conducted under anesthesia. Mild hearing loss: 21-40 decibels hearing level (dBHL), moderate hearing loss: 41-70 dBHL, severe hearing loss: 71-90 dBHL.
Time Frame: Baseline
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
participants
  Right ear, n=11,3 | 11 | 3
  Left ear, n=11,4 | 11 | 4

21. Secondary Outcome: Number of Participants With Mild, Moderate, or Severe Hearing Loss at 6 Months, as Assessed by The Auditory Brain Response (ABR)
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
participants
  Right ear, n=18,4 | 18 | 4
  Left ear, n=18,4 | 18 | 4

22. Secondary Outcome: Number of Participants With Mild, Moderate, or Severe Hearing Loss at 12 Months, as Assessed by The Auditory Brain Response (ABR)
Description: as for outcome 20
Time Frame: 12 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
participants
  Right ear, n=17,4 | 17 | 4
  Left ear, n=17,5 | 17 | 5

23. Secondary Outcome: Number of Participants With Mild, Moderate, or Severe Hearing Loss at End of Study, as Assessed by The Auditory Brain Response (ABR)
Description: as for outcome 20
Time Frame: End of Study (12 months assessment or early termination)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
participants
  Right ear, n=14,4 | 14 | 4
  Left ear, n=15,4 | 15 | 4

24. Secondary Outcome: Percent of Participants With Profound Hearing Loss, as Assessed by the Auditory Brainstem Response (ABR)
Description: Hearing loss in subjects with MPS IIIA was characterized by assessing the ABR. The ABR is a voltage response evoked by acoustic stimuli as sound is processed along the auditory pathway. It consists of electrical signals resulting from the sum of sound-evoked activity along the auditory nerve and brainstem nuclei. The ABR analysis determines the sound intensity at which a neural response first appears (hearing threshold). Other parameters of interest include amplitude (the number of neurons firing), latency (the speed of transmission), interpeak latency (the time between peaks), and interaural latency (the difference in wave V latency between ears). The interpeak latency I-V interval (or central transmission time) is considered the most reliable index of brainstem function. Auditory brainstem response assessments were conducted under anesthesia. Profound hearing loss: 91+ decibels hearing level (dBHL).
Time Frame: Baseline, 6 months, 12 months, End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Baseline, n=11,3 | 0.0 | 0.0
  6 months, n=18,4 | 0.0 | 0.0
  12 months, n=17,4 | 0.0 | 0.0
  End of Study, n=14,4 | 0.0 | 0.0

25. Post Hoc Outcome: Percent of Participants With Thickened Heart Valves as Assessed by Echocardiography (ECG)
Description: ECG allows a non-invasive assessment of cardiac structure, function, and hemodynamics and can provide essential insight into mechanisms of disease and therapeutic benefit.
Time Frame: 12 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Tricuspid Valve, n=18,6 | 5.3 | 0.0
  Pulmonary Valve, n=18,6 | 0.0 | 0.0
  Mitral Valve, n=18,6 | 57.9 | 66.7
  Aortic Valve, n=18,6 | 15.8 | 16.7

26. Post Hoc Outcome: Percent of Participants With Trace Regurgitation as Assessed by ECG
Description: ECG allows a non-invasive assessment of cardiac structure, function, and hemodynamics and can provide essential insight into mechanisms of disease and therapeutic benefit. Regurgitation indicates that blood flows backwards through the valve.
Time Frame: 12 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
percentage of participants
  Tricuspid Valve, n=18,6 | 73.7 | 100.0
  Pulmonary Valve, n=16,5 | 63.2 | 66.7
  Mitral Valve, n=18,6 | 36.8 | 16.7
  Aortic Valve, n=18,6 | 21.1 | 0.0

27. Post Hoc Outcome: Change From Baseline in Tricuspid Valve Regurgitant Velocity
Description: ECG allows a non-invasive assessment of cardiac structure, function, and hemodynamics and can provide essential insight into mechanisms of disease and therapeutic benefit. Backwards blood flow through the tricuspid valve is measured during one heartbeat. A negative value indicates decreased velocity.
Time Frame: Baseline, 6 months, 12 months, End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
meters/second
  6 months, n=2,1 | -0.325 (0.106) | 1.990 (0.0)
  12 months, n=4,2 | -0.013 (0.210) | 1.210 (1.428)
  End of Study, n=3,1 | -0.087 (0.078) | 2.030 (0.0)

28. Post Hoc Outcome: Change From Baseline in The Ratio of Mitral Valve Early Inflow Velocity (E) to Late Inflow Velocity (A)
Description: ECG allows a non-invasive assessment of cardiac structure, function, and hemodynamics and can provide essential insight into mechanisms of disease and therapeutic benefit. Blood flow through the mitral valve is measured during one heartbeat.The E/A ratio measures the relationship between early (E) and late (A) inflow velocity by dividing E by A. A positive value indicates that either early flow through the mitral valve (E) increased or late flow through the valve (A) decreased.
Time Frame: Baseline, 6 months, 12 months, End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: quotient of E/A
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
quotient of E/A
  6 months, n=4,1 | 0.196 (0.418) | 0.059 (0.0)
  12 months, n=3,1 | 0.293 (0.404) | -0.608 (0.0)
  End of Study, n=4,2 | -0.081 (0.529) | -0.226 (0.096)

29. Post Hoc Outcome: Change From Baseline in Liver Volume as Assessed by Abdominal Magnetic Resonance Imaging (MRI)
Description: Liver volume was obtained via abdominal MRI. A negative value indicates that volume decreased.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
milliliters
  6 months, n=5,2 | 93.00 (237.960) | 190.00 (91.924)
  12 months, n=5,2 | 39.20 (248.532) | 280.00 (32.527)
  End of Study, n=4,2 | 356.00 (197.985) | 188.50 (41.719)

30. Post Hoc Outcome: Change From Baseline in Spleen Volume as Assessed by Abdominal Magnetic Resonance Imaging (MRI)
Description: Spleen volume was assessed via abdominal MRI. A negative value indicates that volume decreased.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
milliliters
  6 months, n=5,2 | 29.60 (63.552) | 11.50 (0.707)
  12 months, n=5,2 | 238.40 (473.682) | 44.00 (2.828)
  End of Study, n=4,2 | 128.50 (71.276) | 13.00 (28.284)

31. Secondary Outcome: Number of Participants With "Somewhat" or "Much" Worse Change in Health as Assessed by The Child Health Questionnaire Parent Form 50 (CHQ-PF50)
Description: The parent form, CHQ-PF50, is designed to measure the physical and psychosocial well-being of children 5 years and older. In this trial it was used to assess the health of children 5 to 18 years of age. It consists of 13 health concepts including 11 multi-item and 2 single-item scales: physical function, role/social-emotional/behavioral, role/social-physical, bodily pain, general behavior, mental health, self-esteem, general health perceptions, change in health, parental impact-emotional, parental impact-time, family activities, and family cohesion. The parental impact scales capture the amount of emotional distress and time limitation experienced by the parent due to the child's physical health, emotional well-being, attention/learning abilities, ability to get along with others, and general behavior. The Change in Health section assesses changes in health over the previous year.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
participants
  Baseline, n=6,4 | 1 | 2
  6 months, n=3,5 | 1 | 1
  12 months, n=7,5 | 3 | 1
  End of Study, n=11,6 | 2 | 3

32. Secondary Outcome: Change From Baseline in The Infant Toddler Quality of Life Questionnaire (ITQoL) Growth And Development Subscale
Description: The ITQoL Questionnaire is a generic, validated health status measure for children aged 2 months up to 5 years, including items and scales to measure aspects of physical functioning, development, pain, mood, behavior, general health, and impact on parents. In this study the ITQoL was also administered to patients who were developmentally functioning at or below the age of years. Growth and development is one of 12 health concepts measured by ITQoL. Transformed scores for all subscales range from 0 to 100, with a higher score indicating better health. A positive value indicates improvement.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
units on a scale
  6 months, n=10 | -8.50 (12.813) | NA (NA) — This scale is not used with children in this age group.
  12 months, n=9 | -20.56 (16.853) | NA (NA) — This scale is not used with children in this age group.
  End of Study, n=4 | -28.13 (13.901) | NA (NA) — This scale is not used with children in this age group.

33. Secondary Outcome: Change From Baseline in The Total Sleep Disturbance (TSD) Score of The Children's Sleep Habits Questionnaire (CSHQ)
Description: The CSHQ is a validated, retrospective, parent-reported sleep screening tool. The questionnaire consists of 35 items that yield a TSD score, as well as 8 subscale scores, including bedtime resistance, sleep duration, parasomnias, sleep disordered breathing, night wakings, daytime sleepiness, sleep anxiety, and sleep onset delay. The questionnaire was designed for children aged 4 to 12 years. Parents were asked to think of a recent "typical" week of their child's sleep and to indicate how often sleep disturbance behaviors occurred. A 3-point scale was used for rating: "usually" if the sleep behavior occurs 5 to 7 times per week, "sometimes" for 2 to 4 times per week, and "rarely" for once or not at all during the week. The TSD score, which is the sum of all responses, included all items of the 8 subscales, but consisted of only 33 items because two on the bedtime resistance and sleep anxiety subscales were identical (range: 0, 99). A negative value indicates less sleep disturbance.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children < 6 Years Old | Children ≥ 6 Years Old
Number analyzed (Participants) | 19 | 6
units on a scale
  6 months, n=8,3 | 1.75 (9.968) | 3.33 (8.145)
  12 months, n=8,3 | -0.13 (9.862) | -2.00 (1.732)
  End of Study, n=7,3 | 0.86 (16.098) | 0.33 (6.028)

34. Other Pre Specified Outcome: Change From Baseline in Total Tau Levels in Cerebrospinal Fluid (CSF)
Description: Tau proteins are involved in the building and stabilization of axonal microtubules in the CNS. The phosphorylation of tau proteins associated with microtubules is believed to be involved in destabilizing axons and extensively phosphorylated tau (ptau) has been observed in patients with Alzheimer disease and other neurodegenerative diseases. Because MPS IIIA is a neurodegenerative disease, CSF tau levels were determined to evaluate the potential role of this process in the natural history of the disease. A negative value indicates that total tau levels decreased.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
picograms/milliliter
  6 months, n=17,6 | -88.9 (236.58) | 54.8 (177.63)
  12 months, n=18,6 | -95.8 (375.45) | -79.8 (96.01)
  End of Study, n=14,5 | -80.9 (562.50) | -133.2 (141.82)

35. Other Pre Specified Outcome: Change From Baseline in Phosphorylated Tau Levels in Cerebrospinal Fluid (CSF)
Description: Tau proteins are involved in the building and stabilization of axonal microtubules in the CNS. The phosphorylation of tau proteins associated with microtubules is believed to be involved in destabilizing axons and extensively phosphorylated tau (ptau) has been observed in patients with Alzheimer disease and other neurodegenerative diseases. Because MPS IIIA is a neurodegenerative disease, CSF phosphorylated tau levels were determined to evaluate the potential role of this process in the natural history of the disease. A negative value indicates that phosphorylated tau levels decreased.
Time Frame: Baseline, 6 months, 12 months, and End of Study (Month 24 assessment or early termination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/milliliter
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Number analyzed (Participants) | 19 | 6
picograms/milliliter
  6 months, n=17,5 | -5.42 (20.722) | -1.56 (6.518)
  12 months, n=18,5 | -15.04 (25.550) | -5.42 (5.508)
  End of Study, n=14,4 | -29.98 (41.190) | -29.45 (9.963)

ADVERSE EVENTS:
Groups:
- Children < 6 Years: Patients ≥1 to < 6 years of age with MPS IIIA who were untreated with any investigational products (drugs and/or devices).
- Children ≥ 6 Years: Patients ≥ 6 years of age with MPS IIIA who were untreated with any investigational products (drugs and/or devices).
Arm/Group | Children < 6 Years | Children ≥ 6 Years
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/6
Other Adverse Events (participants affected / at risk) | 8/19 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children < 6 Years (N=19) | Children ≥ 6 Years (N=6)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Ear Haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information (excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication.